CLINICAL TRIAL: NCT01454544
Title: A One Year Trial Evaluating the Safety and Efficacy of the ALK House Dust Mite Allergy Tablet
Acronym: MT-06
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ALK-Abelló A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MT-06; 2011-002277-38 (EudraCT Number)
Record Dates: First submitted 2011-10-13; First posted 2011-10-19 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2017-01

CONDITIONS: House Dust Mite Allergy
MeSH Terms: conditions — Dust Mite Allergy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- ALK house dust mite tablet 6 DU (Experimental)
  Interventions: Biological: AIT Tablet
- ALK house dust mite tablet 12 DU (Experimental)
  Interventions: Biological: AIT Tablet
- Placebo (Placebo Comparator)
  Interventions: Biological: AIT Tablet

INTERVENTIONS:
Biological: AIT Tablet — 1 tablet per day in 12 months

SUMMARY:
The primary aim of this trial is to evaluate the efficacy of the ALK house dust mite tablet given once daily compared to a placebo tablet in the treatment of house dut mite allergic rhinits.

Additionally the secondary objective of the trial is to evaluate the safety and tolarability of the ALK house dust mite tablet.

Immunotherapy has been shown to provide therapeutic benefits to subjects with house dust mite induced allergy. This trial is planned to investigate if clinically relevant improvements in rhinitis symptoms and with less use of symptomatic medication can be obtained in subjects with a history of poor didease control despite of use of symptomatic medications.

ELIGIBILITY:
Inclusion Criteria:

* A history of house dust mite allergy
* Use of symptomatice medication for treatment of house dust mite allergy
* Positive skin prick test to mites
* Positive specific IgE

Exclusion Criteria:

* History of uncontrolled asthma
* Overlapping symptomatice allergies
* Previous treatment with immunotherapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 992 (Actual)
Dates: Start 2011-10; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Evaluation of allergy symptoms and use of symptomatic medication | 1 year with treatment
  Comparing the daily recording of symptoms and use of symptomatic medication during the last period of the trial between the actively treated patients and the placebo treated.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Respiratory Diseases, Lapeyronie Hospital, Montpellier, Montpellier, France

REFERENCES:
- [Derived] Bernstein DI, Kleine-Tebbe J, Nelson HS, Bardelas JA Jr, Sussman GL, Lu S, Rehm D, Svanholm Fogh B, Nolte H. SQ house dust mite sublingual immunotherapy tablet subgroup efficacy and local application site reaction duration. Ann Allergy Asthma Immunol. 2018 Jul;121(1):105-110. doi: 10.1016/j.anai.2018.04.007. Epub 2018 Apr 12. PMID 29656145
- See also: SQ house dust mite (HDM) SLIT-tablet provides clinical improvement in HDM-induced allergic rhinitis — http://www.ncbi.nlm.nih.gov/pubmed/26788764